CLINICAL TRIAL: NCT07225907
Title: Education and Safety for Children With Autism to Prevent Elopement (ESCAPE) Kits Study
Brief Title: ESCAPE Kits for Elopement Prevention in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00108386
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Child Safety; Caregiver Stress
Keywords: Autism Spectrum Disorder; Elopement Behavior; Behavioral Safety Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESCAPE Kits Intervention (Experimental): Family received elopement prevention kits at no cost to them
  Interventions: Behavioral: Elopement Prevention Kits

INTERVENTIONS:
Behavioral: Elopement Prevention Kits — Kits included high locks / bolts on doors (Wideskall 3" gate door latch), door/window alarm (GE 45117 Wireless Alarm with Programmable Keypad), stop sign visual aid (reusable sticker from stickergenius.com), ID tag (SmartKidsID Child ID / Medical ID shoe tag), Bluetooth tracker (BzT patch), safety harness (Dr. Meter AntiLost Link), temporary tattoos (SafetyTat), an information sheet that includes a disclaimer that kit items should be used as intended by manufacturer, that caregivers should monitor the continued proper use of kit items, and that the use of kit items is not a substitute for proper adult supervision of the child. This sheet also included other commonly-recommended EPM such inclusion of elopement accommodations in the child's individualized education plan (if applicable), informing neighbors and/or local law enforcement about the child's elopement behavior, use of safety gates at home, use of temporary tattoos, social stories, and consideration for swimming lessons.

SUMMARY:
This study will evaluate elopement prevention kits for children with autism spectrum disorder who exhibit elopement behavior such as dashing or wandering away from safe settings. Caregivers will be asked to rate how useful individual kit items are at reducing elopement, and to provide feedback about how ESCAPE kits affect their stress levels and ability to engage meaningfully in community settings. This study will also investigate how useful kit items are for various age groups in childhood and adolescence. Information will be used to guide development of a larger elopement prevention program.

DETAILED DESCRIPTION:
open-label feasibility study evaluates the ESCAPE elopement prevention kits for children with autism spectrum disorder (ASD). Kits include safety tools and visual aids intended to reduce elopement behavior. Caregivers assess the usefulness of each item and report on continued use, stress levels, and perceived impact on elopement behavior. Data will inform future large-scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children ages 4-11 years old with a formal diagnosis of ASD (per caregiver report) who have contacted the study team expressing concerns regarding elopement behavior.

Exclusion Criteria:

* Participant doesn't live with the child.
* Only one child under the participant's care can receive the kit.
* Participant doesn't confirm their name, mailing address, and preferred email for kit delivery and post-intervention survey reception.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Kit Items Still in Use at 3 Months | 3 months after kit reception
  Count of individual ESCAPE kit items still actively used by caregivers, reported via REDCap survey.
Caregiver-Rated Usefulness of Individual Kit Items | 3 months after kit reception
  Caregiver ratings of each ESCAPE kit item using a 5-point Likert scale (1 = Not Useful to 5 = Extremely Useful), collected via REDCap survey 3 months post-kit distribution

SECONDARY OUTCOMES:
Caregiver Perception of Kit Impact | 3 months after kit reception
  Caregiver report of impact of kit on the child's elopement, caregiver's personal stress related to child's elopement behavior, and financial burden in having received kit items at no cost to them.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Pereira-Smith, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States